CLINICAL TRIAL: NCT04804917
Title: Long-term Outcome of a Transdiagnostic Cognitive-behavioral Psychotherapy Compared With Management as Usual for Youth With Common Mental Health Problems: a 3-year Follow-up of a Randomized Clinical Trial
Brief Title: 3-year Follow-up of the Mind My Mind RCT
Acronym: MindMyMindFU
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Frederiksberg University Hospital (Other); Defactum, Central Denmark Region (Other Government); The Danish Mental Health Foundation (Other)
Responsible Party: Principal Investigator, Pia Jeppesen, MD, Associate clinical professor, PhD,, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Other Study IDs: MHSCRDenmark, F-61502-03-1
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Emotional Problem; Anxiety Disorder of Childhood; Depressive Symptoms; Behavior Problem of Childhood and Adolescence; Mental Health Disorder
Keywords: Cognitive Behavioral Therapy; Long-term follow-up of RCT; Effectiveness; Transdiagnostic; Children; Adolescents; Youths; Indicated prevention; Personalized treatment
MeSH Terms: conditions — Depression; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants in the MindMyMind RCT: The study participants comprise the 396 youths (and their parents) who participated in the Mind My Mind RCT. The study participants were randomized to the experimental MMM intervention (n=197) or MAU (n=199) and followed in the trial until 26 weeks after randomization, from September 7, 2017, to August 28, 2019.
  The MMM consisted of 9-13 weekly, individual therapy sessions. The CBT methods were organized in modules for anxiety, depression and behavioral problems. Flowcharts described the sequencing and dosing of modules to match the problems at hand. The therapy was completed within 17 weeks, followed by a booster session after four weeks.
  The MAU was enhanced by two care-coordination visits (week 2 and 17). The MAU interventions included anonymous counseling, pedagogical advice, network meetings, educational support, psychological treatment, or no treatment.

SUMMARY:
This is a three-year follow up of a previously completed randomized clinical trial (RCT) of a transdiagnostic cognitive and behavioral (CBT) program ("Mind My Mind" [MMM]) compared to management as usual (MAU) in youth with emotional and behavioral problems.

The effectiveness trial (Clinical Trials Identifier: NCT03535805) evaluated an intervention for help-seeking youth with emotional and behavioral health problems below the threshold for referral to specialized treatment. The experimental intervention MMM consisted of 9-13 weekly, individual therapy sessions delivered by psychologists in a non-specialist school-based setting. The CBT-methods were organized in modules for anxiety, depression and/or behavioral problems, and the therapy was completed within 17 weeks. The MAU was enhanced by two care-coordination visits to help coordinate the usual care in the four municipalities in Denmark. The trial was conducted in four diverse municipalities in Denmark.

The aim of this study is to determine the long-term effects of the transdiagnostic, modular CBT program ("Mind My Mind" [MMM]) compared to management as usual (MAU).

The three-year follow-up of the RCT of MMM versus MAU is nested in a larger study of help-seeking youth screened for eligibility and stratified into three groups with increasing severity of problems. Youths with an intermediate level of problems were included in the RCT. We screened 573 help-seeking youths, and we included and randomized a total of 396 youths (age 6-16 years, with anxiety, depressive symptoms, and/or behavioral problems) to MMM (n=197) or MAU (n=199).

The study participants comprise the 396 youths and their parents who participated in the RCT. We will use the help-seeking population and the background population in the four municipalities as reference groups.

The follow-up study does not include an intervention. The long-term outcome of MMM versus MAU will be investigated using parent-reported questionnaires administered in average three years after random allocation to intervention. All study participants are followed in the Danish national registries.

DETAILED DESCRIPTION:
Background: Behavioral and cognitive-behavioral therapy (CBT) programs targeting a single class of problems are effective, however, these interventions have not been widely implemented, and the population of youth with common mental health problems is markedly undertreated. This knowledge-practice gap calls for pragmatic trials testing the long-term effectiveness of scalable interventions for common mental health problems among youth.

Objective: This is a three-year follow up of a previously completed, randomized clinical trial (RCT) of a transdiagnostic cognitive and behavioral (CBT) program ("Mind My Mind" [MMM]) compared to management as usual (MAU) in youth with emotional and behavioral problems. The RCT (Clinical Trials Identifier: NCT03535805) evaluated a scalable, transdiagnostic intervention for help-seeking youth with emotional and behavioral health problems below the threshold for referral to specialized mental health services.

The specific aim of this follow-up study is to determine the long-term effects of the transdiagnostic and modular CBT program ("Mind My Mind" [MMM]) compared to management as usual (MAU). The secondary aim is to conduct a cost-effectiveness analysis of MMM versus MAU.

Design: This long-term follow-up of the MMM versus MAU is nested in a larger observational study of the population of help-seeking youths who were screened for eligibility. We used a stage-based approach to identify youths with mental health problems requiring an intervention and to stratify the youths into three groups with increasing severity of problems. The youth with an intermediate level of emotional and behavioral problems were included in the RCT. The long-term outcome of the two comparison groups in the RCT will be investigated by administration of research questionnaires to the parents, and the total study population will be described by use of register-based data. The combined use of questionnaires and register-based data will minimize problems of attrition.

Setting: Non-specialist school-based settings in four municipalities in Denmark.

Participants: In summary, 573 help-seeking youths (age 6-16 years) and their parents took part in the screening. Seventy-five (13%) had mental health problems below the intervention threshold, 396 (69%) were deemed eligible for the early intervention and included in the RCT, and 52 (9%) had symptoms of severe mental health problems and disorders and were referred to specialized services. Fifty (9%) youth were excluded for other reasons. A total of 396 youths were identified with anxiety, depressive symptoms, and/or behavioral disturbances. This group was included in the RCT and randomized to MMM (n=197) or MAU (n=199). The primary outcome was the impact of mental health problems reported by the parent at week 18, using the Strengths and Difficulties Questionnaire (SDQ) impact scale (range=0-10 points).

The study participants comprise the 396 youths and their parents who participated in the RCT. We will use the help-seeking population and the background population in the four municipalities as reference groups.

Interventions: The follow-up study does not include an intervention. The MMM consisted of 9-13 weekly, individual therapy sessions delivered by local psychologists who received education and weekly supervision in the MMM manual. The CBT methods were organized in modules for anxiety, depression and behavioral problems. Flowcharts described the sequencing and dosing of modules to match the problems at hand, e.g. parent management training for youth's behavioral problems. The therapy was completed within 17 weeks, followed by a booster session after four weeks.

The MAU was enhanced by two care-coordination visits (week 2 and 17) to help access care in the municipality. The MAU interventions included anonymous counseling, pedagogical advice, network meetings, educational support, private or publicly funded psychological treatment, or no treatment.

Outcomes: The long-term outcome of MMM versus MAU will be investigated using parent-reported questionnaires administered in average three years after random allocation to intervention. All study participants are followed in the Danish national registries by linking of individual-level data from several registries. The follow-up will be conducted approximately three years (30-43 months) after the random allocation to intervention in the RCT.

The register-based exploratory outcomes will focus on the youth's use of psychiatric and somatic health care services, academic performance on the national school tests and exams, school absence and wellbeing in school. Regarding use of health care services, we will study the time to the first contact, and the frequency and the pattern of contacts (acute/non-acute, inpatient/outpatient, psychiatric/somatic) during the follow-up period. We will also track activities in the social sector including notifications to the authorities stating a concern for the health and wellbeing of the young person, and preventative interventions to assist the family. Finally, we will study changes in the parents' employment status (including sick leave, part-time work and unemployment) during the follow-up period to assess whether the participation in MMM, relatively to MAU, did influence the life circumstances of the family in a broader sense.

Cost-effectiveness analysis: The evaluation of the cost-effectiveness of the MMM, relative to MAU, will build on our previous cost-utility analysis (CUA) of data from the RCT. The extended follow-up time will reduce the uncertainty around the results by replacing the extrapolation scenarios with repeated assessment of the health-related quality of life measured with the parent-reported questionnaire CHU9D. The analyses of costs will include register-based, individual-level data on the young person's health care utilization in the 3-year follow-up period from the date of randomization, along with the associated unit costs that are listed in administrative registers.

Perspectives: The study will provide new knowledge of the long-term effectiveness of transdiagnostic CBT to lower the burden of mental health disorders in youth.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the Mind My Mind RCT (n=396)
2. Written consent by the parent and legal guardian to take part in the 3-year follow-up of the Mind My Mind RCT by answering the web-based questionnaires

Exclusion Criteria:

1) Withdrawal from the follow-up of Mind My Mind RCT (n=63).

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study subjects are the 396 school-aged youths who were identified with indicated need for treatment of anxiety, depressive symptoms, and/or behavioral disturbances and randomized to MMM (n=197) or MAU (n=199).
  The parent of each of subject will be invited to answer questionnaires to assess the long-term outcomes.
  We will also follow the help-seeking population (n=573) and the age-matched background population in the four municipalities (study sites) by use of data drawn from the Danish National Registries (reference groups).
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
The child's impact of mental health problems reported by the parent on the Strengths and Difficulties Questionnaire Impact Scale. | Last month at 3-year follow-up
  The parent-reported Strengths and Difficulties Questionnaire (SDQ) Impact Scale is scored from 0 to 10 (1, 2, 3, 4, 5, 6, 7, 8, 9, 10) with higher scores indicating more impact of mental health problems.
  The minimum relevant difference in impact of mental health problems measured by the SDQ Impact Scale was set at 1.0 corresponding to a change from severe to moderate, or from moderate to little-or-no impact in one of the five domains of child's life (distress, home-life, friendships, classroom learning and leisure activities). The SDQ Impact was previously measured at week 0, 2, 4, 6, 8, 10, 12, 14, 18 and 26 asking about the last six months at baseline and asking about the last month at each follow-up.

SECONDARY OUTCOMES:
Emotional and behavioral problems | Last month at 3-year follow-up
  The SDQ contains 25 items, each scored on a 3-point Likert scale (0, 1, 2), and divided into five sub-scales measuring emotional problems, behavioral problems, hyperactivity, peer problems and pro-social behavior. The total difficulties scale consists of 20 items, and the sum is calculated (range 0-40) to measure the emotional and behavioral difficulties across the first four problem areas. Higher scores indicate more severity of problems. The parent-reported total difficulties score was measured at week 0, 18 and 26 asking about the last six months at baseline and asking about the last month at week 18 and 26.
School attendance: proportion of school-days within the last 4 weeks, where the child is present (no illegal absence) | Last four weeks at 3-year follow-up
  Parent reported measures of different kinds of school absence
Child Health Utility instrument (CHU9D) | The present day at 3-year follow-up
  The Child Health Utility instrument (CHU9D) measures the health-related quality of life (QoL) in nine domains. The measure is developed specifically for use among children and adolescents. The CHU9D has nine items with five levels of severity in the domains: worried, sad, pain, tired, annoyed, schoolwork/homework, sleep, daily routine and activities. The raw scores range from 9 to 35, with 9 indicating the highest possible QoL and 35 indicating the poorest QoL. The scores can be converted to utilities ranging 0-1 on the dead-full health QALY scale, using preference-based scoring algorithms. The CHU9D is a validated measure of health-related quality of life for use in youth mental health trials.
  The parent-reported CHU9D was previously measured at week 0, 18 and 26 asking about the present day.
The Parental Stress Scale (PSS) | Present time at 3-year follow-up
  The Parental Stress Scale (PSS) is a parent-reported questionnaire with 18 items, scored on a five-point scale (strongly disagree =1, disagree=2, disagree or agree=3, agree=4, strongly agree=5) for each of the eight positively and ten negatively worded items. The scores of the eight positive items are reversed when coding the PSS, and a single parental stress sum is calculated (range 0-72) with higher scores indicating more parental stress. The PSS measures the stress a parent experiences in the role functioning as parent. The instrument has been validated in Denmark.
  The PSS score was measured at week 0, 18 and 26 asking the parent of the present time (no explicit time frame)

OTHER OUTCOMES:
The number of participants who responded defined as a SDQ Impact score reduction ≥1 points | at 3-year follow-up
  Response was defined as a one-point reduction on the parent-reported impact scale from baseline to follow-up
The number of participants in remission defined as SDQ algorithm scores below cut-off for need of treatment | at 3-year follow-up
  To define the threshold for a child's need of treatment (inclusion in the RCT) we developed and validated the following SDQ algorithm: parent-reported SDQ total-difficulties score ≥14, emotional problems ≥5, and/or conduct score ≥3; combined with a functional impairment score ≥1. This algorithm defined the cut-off for problems above the 90-percentile of mental health problems in the general age-matched population.
  Remission was defined as SDQ-algorithm scores below the threshold that indicate need of treatment.
Psychosocial treatments | Last three months at 3-year follow-up
  Parent-reported questionnaire about the psychosocial treatment and support that their child received in the school-, social-, health-, and private sectors.
The impact of child's mental health problems on the parent's ability to work | Last four weeks at 3-year follow-up
  Parent-reported questionnaire about managing their own obligations at work or in an education, eg arriving late, going home early, taking sick leave.
Parent-reported unmet needs | Present time at 3-year follow-up
  Parent-reported questionnaire about the current mental health problems and unmet needs of their child.
Use of health care services | Time period from randomization to June 30, 2021
  Individual-level data retrieved from the Danish National Patient Register containing information about contacts with the health care system during the follow-up period. Data is collected routinely in the Danish health care system, independent of the present study. Contacts with the health care system will be assessed and compared as incidence rates of acute/non-acute, in-patient/outpatient and psychiatric/somatic contacts.
Use of psychotropic drugs | Time period from randomization to June 30, 2021
  Individual-level data retrieved from the Danish National Drug Database containing information about redeemed prescriptions. Data is collected routinely and independent of this study. Incident use and duration of use of the following psychotropic drugs described by ATC codes (including subgroups contained in the codes) will be studied: C02AC02, N03AE, N05A, N05BA, N05CH, N06A, N06BA, N05CF.
School attendance | Time period from end of intervention (week 18) to June 30, 2021
  Individual-level data retrieved from the Danish Ministry of Education. Data is collected routinely and independent of this study. School attendance consists of several factors: a) the type of schooling that the child/youth is currently attending, and b) the frequency and proportion of school time the child/youth is registered as not attending. The data quality will be affected by the Covid-19 pandemic school shutdowns, meaning that we may have to omit this outcome.
School performance | Time period from end of intervention (week 18) to June 30, 2021
  Individual-level data retrieved from the Danish Ministry of Education. Data is collected routinely and independent of this study. Scores from either a national test of academic performance in Danish or mathematics (one offered at most levels in primary school) in the follow-up period. The score will be assessed with external reference (e. g. national average) as well as relatively among their own peers (e. g. scores divided in tertiles/quartiles). Also, available information on non-attendance at the school tests and exams is considered a relevant outcome, assessed as a frequency and proportional outcome. The data quality will be affected by the Covid-19 pandemic school shutdowns, meaning that we may have to omit this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jeppesen, PhD, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Services in the Capital Region, Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The pseudonymous individual participant data can be made available to investigators for individual participant data meta-analyses that have been approved by independent review committees. The data access will be granted on a case-by-case basis by the principal investigator (Pia Jeppesen) after further approval by the nongovernmental organization Psykiatrifonden (who was responsible for the implementation of the MMM program in the municipalities and has the legal responsibility as the data controller for the Web-based data collection). Access will be granted to the extent permissible by the General Data Protection Regulation and the Danish Data Protection Act. Making the data available may require approval from the Danish Data Protection Authority.

REFERENCES:
- [Result] Jeppesen P, Wolf RT, Nielsen SM, Christensen R, Plessen KJ, Bilenberg N, Thomsen PH, Thastum M, Neumer SP, Puggaard LB, Agner Pedersen MM, Pagsberg AK, Silverman WK, Correll CU. Effectiveness of Transdiagnostic Cognitive-Behavioral Psychotherapy Compared With Management as Usual for Youth With Common Mental Health Problems: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Mar 1;78(3):250-260. doi: 10.1001/jamapsychiatry.2020.4045. PMID 33355633
- [Result] Wolf RT, Puggaard LB, Pedersen MMA, Pagsberg AK, Silverman WK, Correll CU, Plessen KJ, Neumer SP, Gyrd-Hansen D, Thastum M, Bilenberg N, Thomsen PH, Jeppesen P. Systematic identification and stratification of help-seeking school-aged youth with mental health problems: a novel approach to stage-based stepped-care. Eur Child Adolesc Psychiatry. 2022 May;31(5):781-793. doi: 10.1007/s00787-021-01718-5. Epub 2021 Jan 18. PMID 33459884
- [Result] Wolf RT, Ratcliffe J, Chen G, Jeppesen P. The longitudinal validity of proxy-reported CHU9D. Qual Life Res. 2021 Jun;30(6):1747-1756. doi: 10.1007/s11136-021-02774-9. Epub 2021 Feb 13. PMID 33582966